CLINICAL TRIAL: NCT00058266
Title: A Phase II Study Of Genistein In Patients With Localized Prostate Cancer (Molecular Correlates of Soy In Humans)
Brief Title: Genistein in Treating Patients With Localized Prostate Cancer Who Are Planning to Undergo Radical Prostatectomy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Data Monitoring Committee cited poor accrual.
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NU 00U7; NU-00U7
Record Dates: First submitted 2003-04-07; First posted 2003-04-09 (Estimated); Last update posted 2012-07-19 (Estimated); Status verified 2012-07

CONDITIONS: Prostate Cancer
Keywords: stage I prostate cancer; stage II prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Genistein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Experimental): Patients receive oral genistein once daily for 1-2 months, undergo radical prostatectomy, and then continue oral genistein once daily for 1-2 months afterward (for a total of 3 months of therapy).
  Interventions: Dietary Supplement: genistein; Procedure: conventional surgery
- Group B (Experimental): Patients undergo radical prostatectomy. Beginning 1 month after surgery, patients receive genistein as in arm I for 3 months.
  Interventions: Dietary Supplement: genistein; Procedure: conventional surgery

INTERVENTIONS:
Dietary Supplement: genistein — Given orally
Procedure: conventional surgery — Patients undergo surgery

SUMMARY:
RATIONALE: Genistein may stop the growth of cancer cells by blocking the enzymes necessary for cancer cell growth.

PURPOSE: Phase II trial to study the effectiveness of genistein in treating patients with localized prostate cancer who are planning to undergo radical prostatectomy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the toxicity of genistein in patients with localized prostate cancer treated with radical prostatectomy.
* Determine the decrease, if any, of prostate-specific antigen-positive cells in the operative field of patients treated with this drug.
* Determine the quality of life of patients treated with this drug.

OUTLINE: Patients receive 1 of 2 treatment regimens.

* Group A: Patients receive oral genistein once daily for 1-2 months, undergo radical prostatectomy, and then continue oral genistein once daily for 1-2 months afterward (for a total of 3 months of therapy).
* Group B: Patients undergo radical prostatectomy. Beginning 1 month after surgery, patients receive genistein as in arm I for 3 months.

Quality of life is assessed at baseline and at 1 and 3 months after surgery.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 88 patients (44 patients per treatment group) will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of localized prostate cancer

  * Diagnosed within the past 6 months
  * T1 or T2 disease
  * Gleason score 5-8
  * Prostate-specific antigen no greater than 20 ng/mL
* Radical prostatectomy planned

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-1

Life expectancy

* More than 2 years

Hematopoietic

* Hemoglobin greater than 9.0 g/dL
* Platelet count greater than 100,000/mm^3
* Absolute neutrophil count greater than 1,000/mm^3

Hepatic

* SGPT and SGOT less than 3 times normal
* Bilirubin less than 3 mg/dL (less than 1.5 times normal) (patients with an elevated bilirubin due to a familial defect in bilirubin metabolism will be considered on an individual basis)

Renal

* Creatinine less than 2.0 mg/dL

Cardiovascular

* No venous thrombosis within the past year

Other

* Patients must use effective barrier contraception
* No other medical condition that would preclude study therapy
* No known soy intolerance

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* No concurrent hormonal therapy for prostate cancer

Radiotherapy

* Not specified

Surgery

* See Disease Characteristics

Other

* No concurrent soy supplements
* No concurrent foods high in genistein
* No concurrent active therapy for neoplastic disorders

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2002-12; Primary Completion 2006-11 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Toxicity | At surgery & monthly thereafter during treatment (3 mos)
Decrease in prostate-specific antigen-positive cells | At time of surgery
Alteration in cell morphology | At time of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Raymond C. Bergan, MD, Study Chair — Robert H. Lurie Cancer Center
Locations (5):
- United States (5):
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Veterans Affairs Medical Center - Lakeside Chicago, Chicago, Illinois
  - Evanston Northwestern Healthcare - Evanston Hospital, Evanston, Illinois
  - Ingalls Cancer Care Center at Ingalls Memorial Hospital, Harvey, Illinois
  - University of Washington School of Medicine, Seattle, Washington